CLINICAL TRIAL: NCT03697343
Title: Efficacy and Safety of Fractionated Stereotactic Radiotherapy (FSRT) in Comparison to Single Session Radiosurgery in Patients With Larger Brain Metastases (2-4 cm)
Brief Title: Fractionated Stereotactic Radiotherapy vs. Single Session Radiosurgery in Patients With Larger Brain Metastases
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSRT-Trial
Record Dates: First submitted 2018-09-26; First posted 2018-10-05 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Cerebral Metastases of Solid Cancers
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, Open-Label, randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiosurgery with 1 x 18 Gy (2-3 cm) or 1 x 15 Gy (3-4 cm) and (Other): Radiosurgery with 1 x 18 Gy (2-3 cm) or 1 x 15 Gy (3-4 cm) and no margin as defined by the RTOG 9005
  Interventions: Radiation: Radiosurgery
- Fractionated stereotactic radiotherapy with 12 x 4 Gy and 2 mm (Other): Fractionated stereotactic radiotherapy with 12 x 4 Gy and 2 mm margin
  Interventions: Radiation: Fractionated stereotactic radiotherapy

INTERVENTIONS:
Radiation: Radiosurgery — Radiosurgery with 1 x 18 Gy (2-3 cm) or 1 x 15 Gy (3-4 cm)
  Arms: Radiosurgery with 1 x 18 Gy (2-3 cm) or 1 x 15 Gy (3-4 cm) and
Radiation: Fractionated stereotactic radiotherapy — Fractionated stereotactic radiotherapy with 12 x 4 Gy and 2 mm
  Arms: Fractionated stereotactic radiotherapy with 12 x 4 Gy and 2 mm

SUMMARY:
Phase III trial comparing local control and side effects after fractionated stereotactic radiotherapy and single session radiosurgery in patients with larger brain metastases (2-4 cm)

DETAILED DESCRIPTION:
This is a prospective, multicenter randomized trial comparing local control and side effects after fractionated stereotactic radiotherapy with 12 x 4 Gy and single session radiosurgery according to RTOG 9005 in patients with larger brain metastases (2-4 cm). Patients will be randomized to either fractionated stereotactic radiotherapy with 12 x 4 Gy or radiosurgery with 1 x 18 Gy (2-3 cm) or 1 x 15 Gy (3-4 cm) as defined by the RTOG 9005. Randomization will be stratified by metastasis volume and histology.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years, no upper age limit
* Karnofsky Performance Score > 50 points
* Expected Survival > 3 months
* 1-10 cerebral metastases of metastatic solid cancer
* Indication for local radiotherapy
* Patients must be able to understand the protocol and provide informed consent

Exclusion Criteria:

* Whole Brain radiotherapy no longer than 6 weeks before the start of stereotactic radiotherapy or planned whole brain radiotherapy after stereotactic radiotherapy
* Prior irradiation of the cerebral metastasis that is to be treated in the study
* Relevant overlap of prior radiation fields with the metastasis that is to be treated in the study
* Metastasis in the brainstem
* Contraindication for cerebral MRI
* Metastasis that is to be treated in the study can't be visualized in contrast-enhanced T1 MRI sequence
* Pregnant or lactating women
* Abuse of illicit drugs, alcohol or medication
* Patient not able or willing to behave according to protocol
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Time to local progression - TTLP | 12 months
  Local progression will be defined according to the RANO-BM criteria by an increase of at least 20% in the longest diameter of the metastasis relative to nadir or baseline. In addition to the relative increase of 20% the lesion must increase by an absolute value of 5 mm or more.
  TTLP is defined as the time from randomization until the detection of progression as per the RANO-BM criteria. Patients will be censored if they have no signs of local progression at the time of last tumor monitoring during follow-up or at the onset of one of the following competing risk events not associated with local progression: death, lost to follow up, unauthorized non-protocol treatment of the target lesion.
  Confirmatory analysis of the primary endpoint variable will be performed using a p-value of p≤0.05 as the global significance level.

SECONDARY OUTCOMES:
CNS toxicity according to CTCAE v5.0 | 12 months
  CNS toxicity according to CTCAE v5.0
Time to local progression (Volumetric RANO-BM criteria) | 12 months
  Based on the RANO-BM criteria, progression is defined as an increase in volume of 72.8% or more (corresponds to a 20% increase in diameter for a perfect sphere).
Quality of Life according to EORTC QLQ-C30 | Change from baseline to 3, 6, 12 and 24 months
  Quality of life measured by European Organization for Research and Treatment of Cancer (EORTC) questionnaire QLQ C30
Local-Progression-Free Survival | 12 months
  Local-Progression-Free Survival is defined like TTLP except that death not associated with local progression will not be censored but assessed as a separate event
Overall Survival | 24 months
  Overall Survival
Quality of Life according to EORTC QLQ-BN20 | Change from baseline to 3, 6, 12 and 24 months
  Quality of life measured by European Organization for Research and Treatment of Cancer (EORTC) questionnaire QLQ BN20

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Fietkau, Prof., Principal Investigator — Universitätsklinikum Erlangen, Strahlenklinik; Florian Putz, PD Dr.med., Principal Investigator — Universitätsklinikum Erlangen, Strahlenklinik
Locations (13):
- Germany (13):
  - Klinik für Strahlentherapie und Radioonkologie Stuttgart, Stuttgart, Baden-Wurttemberg
  - Klinik für Strahlentherapie Bayreuth, Bayreuth, Bavaria
  - Strahlentherapie Coburg, Coburg, Bavaria
  - Radio-Log Strahlentherapie Hof, Hof, Bavaria
  - Strahlentherapie Süd Kempten, Kempten (Allgäu), Bavaria
  - Klinik und Poliklinik für RadioOnkologie und Strahlentherapie München (TUM), München, Bavaria
  - Klinik und Poliklinik für Strahlentherapie Regensburg, Regensburg, Bavaria
  - Klinik für Strahlentherapie und Radioonkologie, Bonn, North Rhine-Westphalia
  - Klink und Praxis für Radioonkologie Chemnitz, Chemnitz, Saxony
  - Universitätsklinik und Poliklinik für Strahlentherapie Halle, Halle, Saxony-Anhalt
  - Klinik für Strahlentherapie und Radioonkologie Universitätsklinikum Jena, Jena, Thuringia
  - Klinik für Radioonkologie und Strahlentherapie Charité Berlin, Berlin
  - Erlangen, Universitätsklinikum Strahlenklinik, Erlangen